CLINICAL TRIAL: NCT05137600
Title: A Phase 1, Open-label, 2-cohort, Fixed-sequence, Drug-drug Interaction Study to Investigate the Potential Interaction Between ATI-2173 When Coadministered With Midazolam or Clarithromycin in Healthy Subjects
Brief Title: A Drug-Drug Interaction Study Between ATI-2173 and Midazolam or Clarithromycin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Antios Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ANTT103
Record Dates: First submitted 2021-10-28; First posted 2021-11-30 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Drug Drug Interaction
MeSH Terms: interventions — Midazolam; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ATI-2173 50 mg (Experimental): ATI-2173 is a liver-targeted phosphoramidate prodrug of clevudine designed to enhance anti-HBV activity while decreasing systemic exposure to clevudine. It will be dosed as a capsule by mouth
  Interventions: Drug: ATI-2173
- Midazolam (Experimental): Midazolam is a sensitive CYP3A index substrate
  Interventions: Drug: Midazolam
- Clarithromycin (Experimental): Clarithromycin is a sensitive P-gp index inhibitor to evaluate potential effect of P-gp inhibition on ATI-2173 and its metabolites
  Interventions: Drug: Clarithromycin

INTERVENTIONS:
Drug: ATI-2173 — ATI-2173 is a liver-targeted phosphoramidate prodrug of clevudine designed to enhance anti-HBV activity while decreasing systemic exposure to clevudine. It will be dosed as a capsule by mouth
  Arms: ATI-2173 50 mg
Drug: Midazolam — Midazolam is a sensitive CYP3A index substrate
  Arms: Midazolam
Drug: Clarithromycin — Clarithromycin is a sensitive P-gp index inhibitor to evaluate potential effect of P-gp inhibition on ATI-2173 and its metabolites(clarithromycin)
  Arms: Clarithromycin

SUMMARY:
This study is a single-center, open-label, 2-cohort, fixed-sequence, DDI study in healthy adult subjects. Healthy volunteers will be administered multiple oral doses of ATI-2173 in combination with midazolam or clarithromycin and assessed for safety and tolerability including blood tests to show how the body metabolizes and eliminates the investigational drug as well as how the investigational drug interacts with midazolam or clarithromycin.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated Informed Consent Form (ICF)
2. Stated willingness to comply with all study procedures (including ability and willingness to abstain from alcohol from 48 hours prior to the first study drug administration until discharge) and availability for the duration of the study
3. Healthy adult male or female
4. Aged between 18 and 60 years, inclusive
5. Body mass index (BMI) within 18.5 kg/m2 to 30.0 kg/m2, inclusively
6. Non- or ex-smoker (an ex-smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first study drug administration)
7. Suitable veins for cannulation or repeated venipuncture as assessed by an Investigator at Screening
8. If female, meets one of the following criteria:

   1. Is of childbearing potential and agrees to use an acceptable contraceptive method. Acceptable contraceptive methods include

      * Abstinence from heterosexual intercourse from the first study drug administration through to at least 60 days after the last dose of the study drug
      * Non-hormonal intrauterine device (IUD) with a barrier method (eg, male condom) used from at least 28 days prior to the first study drug administration through to at least 60 days after the last dose of the study drug
      * Double-barrier method (eg, male condom, spermicide and diaphragm or cervical cap used simultaneously )from Screening through to at least 60 days after the last dose of the study drug
      * Male partner vasectomized at least 6 months prior to Screening Or
   2. Is of non-childbearing potential, defined as surgically sterile (ie, has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or is in a postmenopausal state (ie, at least 1 year without menses without an alternative medical condition prior to the first study drug administration), as confirmed by follicle-stimulating hormone levels (≥ 40 mIU/mL).
9. If male, meets one of the following criteria:

   1. Is able to procreate and agrees to use one of the accepted contraceptive regimens and not to donate sperm from the first study drug administration to at least 90 days after the last drug administration. An acceptable method of contraception includes one of the following:

      * Abstinence from heterosexual intercourse
      * Male condom with spermicide or male condom with a vaginal spermicide (gel, foam, or suppository) Or
   2. Is unable to procreate; defined as surgically sterile (ie, has undergone a vasectomy at least 6 months prior to Screening)
10. Agrees to abstain from blood or plasma donation from the Screening visit until 3 months after the last study drug administration
11. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination, vital signs, myopathy questionnaire, and/or ECG, as determined by an Investigator Cohort 1 only
12. Have no clinically significant findings on the neurological examination and/or oxygen saturation measurement as determined by an Investigator

Exclusion Criteria:

1. Female who is lactating
2. Female who is pregnant according to the pregnancy test at Screening or prior to the first study drug administration
3. Female using the following systemic contraceptives: oral, patch or vaginal ring, in the 28 days prior to the first study drug administration
4. Female using hormone replacement therapy in the 28 days prior to the first study drug administration
5. Female using the following systemic contraceptives: injections or implant, or hormone-releasing IUD in the 13 weeks prior to the first study drug administration
6. Seated pulse rate less than 50 beats per minute or more than 100 beats per minute at Screening or prior to the first study drug administration
7. Seated blood pressure below 105/60 mmHg or higher than 140/90 mmHg at Screening or prior to the first study drug administration
8. Estimated glomerular filtration rate (eGFR) ≤ 60 mL/min/1.73m2, calculated using the Modification of Diet in Renal Disease (MDRD) equation, at Screening or prior to the first study drug administration
9. Presence of out-of-range cardiac interval (PR < 110 msec, PR > 200 msec, QRS < 60 msec, QRS >110 msec and QTcF > 440 msec) on the ECG at Screening or at Check-in or other clinically significant ECG abnormalities, unless deemed non-significant by an Investigator
10. Hemoglobin value below the lower limit of the reference laboratory at Screening or prior to study drug administration
11. Any other clinically significant abnormalities in laboratory test results at Screening. Subjects with alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), creatine kinase (CK) or total bilirubin outside the normal range at Screening or Day -1 will be excluded.
12. Positive test result for alcohol and/or drugs of abuse at Screening or prior to the first drug administration
13. Positive screening results to HIV Ag/Ab combo, hepatitis B surface antigen or hepatitis C virus antibody tests at Screening
14. Positive screening results to SARS-CoV-2 virus tests prior to the first study drug administration
15. History of significant hypersensitivity to ATI-2173, clevudine, midazolam, clarithromycin, or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
16. Presence or history of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability
17. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
18. Presence of clinically significant muscle disorders, myopathies or other forms of liver disease
19. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
20. Any clinically significant illness in the 28 days prior to the first study drug administration
21. Use of any prescription drugs (including hormonal contraceptives and hormone replacement therapy) or any CYP3A inhibitors, inducers, or substrates in the 30 days prior to the first study drug administration, that in the opinion of an Investigator would put into question the status of the participant as healthy
22. Use of St. John's wort in the 30 days prior to the first study drug administration
23. Use of over-the-counter (OTC) medications, herbal supplements, and vitamins in the 14 days prior to the first study treatment administration.
24. Use of quinine-containing products (eg, tonic water), grapefruit products, pomelo products, Seville orange products, including supplements containing Citrus aurantium or "bitter orange", in the 14 days prior to the first study drug administration
25. Consumption of food or beverages containing xanthines (ie, tea, coffee, cola drinks, energy drinks or chocolate) in the 48 hours prior to the first study drug administration
26. Any history of tuberculosis
27. Immunization with a coronaviruse disease 2019 (COVID-19) vaccine in the 14 days prior to the first study drug administration
28. Scheduled immunization with a COVID-19 vaccine (first or second dose) during the study that, in the opinion of an Investigator, could potentially interfere with subject participation, subject safety, study results, or any other reason
29. Inclusion in a previous group for this clinical study
30. Participation in another clinical study with a non-biologic investigational product (IP) or new formulation of a marketed non-biologic drug in the 30 days prior to Screening
31. Participation in another clinical study with any marketed or investigational biologic product within 90 days or 5 half-lives, whichever is longer, prior to Screening
32. Donation of 50 mL or more of blood in the 28 days prior to the first study drug administration
33. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the 56 days prior to the first study drug administration Cohort 1
34. Oxygen saturation (SpO2) below 95% at Screening or prior to the first study drug administration
35. Family history of sudden cardiac death or known prolonged QTc

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2022-01-23 (Actual)

PRIMARY OUTCOMES:
Cmax of Midazolam | Through end of study, approximately 3 months
AUC0-t of Midazolam | Through end of study, approximately 3 months
AUC0-inf of Midazolam | Through end of study, approximately 3 months
Cmax of ATI-2173 | Through end of study, approximately 3 months
AUCtau of ATI-2173 | Through end of study, approximately 3 months
AUC0-t of ATI-2173 | Through end of study, approximately 3 months
AUCo-inf of ATI-2173 | Through end of study, approximately 3 months

SECONDARY OUTCOMES:
Number of adverse events | Through end of study, approximately 3 months

OTHER OUTCOMES:
Cmax of 1-hydroxymidazolam | Through end of study, approximately 3 months
AUC0-t of 1-hydroxymidazolam | Through end of study, approximately 3 months
AUC0-inf of 1-hydroxymidazolam | Through end of study, approximately 3 months
Ratio of metabolite to parent (midazolam) for AUC0-t | Through end of study, approximately 3 months
Ratio of metabolite to parent (ATI-2173) for AUC0-t | Through end of study, approximately 3 months
Ratio of metabolite to parent (ATI-2173) for AUCtau | Through end of study, approximately 3 months
Cmax of M1 | Through end of study, approximately 3 months
AUC0-t of M1 | Through end of study, approximately 3 months
AUC0-inf of M1 | Through end of study, approximately 3 months
Cmax of clevudine | Through end of study, approximately 3 months
AUCtau of clevudine | Through end of study, approximately 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No